CLINICAL TRIAL: NCT03578042
Title: Effect of Fixed Triple Combination With Losartan-Amlodipin-HCTZ vs. Free Triple Combination on Blood Pressure Control
Brief Title: Fixed-Free HTN Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Principal Investigator, Rabih Azar, MD, MPH, Chief of Cardiology, Hotel Dieu de France Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Losanet AM Plus trial
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Amlodipine; Hydrochlorothiazide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LosanetAMplus (Active Comparator): Patients taking the fixed triple combination
  Interventions: Drug: Losartan and amlodipine and hydrochlorothiazide
- standard of care (Other): Patients taking 2 or 3 free combinations containing 3 drugs for hypertension as decided by the treating physician
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Losartan and amlodipine and hydrochlorothiazide — this is a fixed combination containing the 3 drugs
  Arms: LosanetAMplus
Drug: Standard of care — any free triple combination therapy for hypertension given as 2 or 3 pills
  Arms: standard of care

SUMMARY:
Evaluation of the effect of FIXED triple anti-hypertensive therapy with losartan-amlodipin-HCTZ vs any free triple combination therapy chosen by the treating physician for patients with uncontrolled hypertension

DETAILED DESCRIPTION:
Patients who have uncontrolled hypertension and who require triple therapy will be randomized to receive:

1. Fixed combination containing 3 anti-hypertensive drugs: losartan 100 mg + amlodipin 5 mg + hydrocholorothiazide 12.5 mg one tab/day
2. Or any other therapy decided by the treating physician containing three anti-hypertensive agents but supplied as "free" therapy, meaning supplied as 2 or 3 separate tablets Patients will have a baseline ambulatory blood pressure recording. The same recording will be repeated at 2 months of therapy.

We expect fixed triple combination to be more effective because the drugs used work synergistically together and the compliance will be higher

ELIGIBILITY:
Inclusion Criteria:

* Patients already on free triple anti-HTN therapy whether controlled or not Or patients on double anti-HTN therapy who are uncontrolled* Or patients on monotherapy and who have a BP > 160/100 mm Hg

  * BP is defined as UNCONTROLLED if > 135/85 at home or > 140/90 in clinic on at least 2 occasions

Exclusion Criteria:

* Contra-indication for the use of ARB or ACEI, CCB or hydrochlorothiazide History of angina pectoris or myocardial infarction < 3 months old Permanent atrial fibrillation Ejection fraction < 40% Patients with hypertension but who are not on any medication Patients with hypertension and who are treated with > 3 drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
average 24 hour blood pressure measured by ambulatory recording | measured after 2 months of therapy
  Measured by ambulatory blood pressure recording over 24 hours

SECONDARY OUTCOMES:
central aortic blood pressure | measured after 2 months of therapy
pulse wave velocity | measured after 2 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rabih R Azar, MD, MPH, Principal Investigator — Hotel Dieu de France Hospital
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No